CLINICAL TRIAL: NCT00369343
Title: A Multicenter, Randomized, 8-week, Double-blind, Placebo-controlled Study Followed by a 6-month Open-label Extension to Evaluate the Efficacy and Safety of DVS SR in Peri- and Postmenopausal Women With Major Depressive Disorder
Brief Title: Study Evaluating Desvenlafaxine Succinate Sustained Release (DVS SR) Versus Placebo in Peri- and Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3151A1-403
Record Dates: First submitted 2006-08-25; First posted 2006-08-29 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Depression; Depressive Disorder; Depressive Disorder, Major
Keywords: Major Depressive Disorder; vasomotor symptoms; menopause; diabetic neuropathy; fibromyalgia
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major; Diabetic Neuropathies; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Desvenlafaxine administered as a succinate salt in a sustained-release form (DVS SR)
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desvenlafaxine administered as a succinate salt in a sustained-release form (DVS SR) — DVS-SR 50-200mg, daily (QD), tablet form, treatment period up to 34 weeks
  Arms: A
Drug: Placebo — Placebo, daily (QD), tablet form, treatment period up to 8 weeks
  Arms: B

SUMMARY:
Desvenlafaxine succinate (DVS) is a potent and selective serotonin and norepinephrine reuptake inhibitor (SNRI). The sustained-release (SR) formulation, DVS SR, is being studied in the development program for the treatment of major depressive disorder (MDD), for vasomotor symptoms (VMS) associated with menopause, and for pain associated with peripheral diabetic neuropathy, as well as for the treatment of fibromyalgia syndrome. This study will investigate the safety, efficacy, and tolerability of DVS SR in women with MDD who are peri- and postmenopausal.

ELIGIBILITY:
Inclusion Criteria:

* Peri- and postmenopausal women between the ages of 40 and 70 years, inclusive.
* A primary diagnosis of MDD, single or recurrent episode, without psychotic features using the modified International Neuropsychiatric Interview (MINI).
* Montgomery-Asberg Depression Rating Scale (MADRS) total score > or = 22 at the screening and baseline visit.

Exclusion Criteria:

* Use of oral estrogen-, progestin-, androgen-, or Selective Estrogen Receptor Modulator (SERM)-containing drug products 8 weeks before baseline.
* Current (within 12 months) psychoactive substance abuse or dependence (including alcohol), manic episode, post-traumatic stress disorder, obsessive-compulsive disorder, or a lifetime diagnosis of bipolar or psychotic disorder.
* A history or active presence of clinically important medical disease.

Additional criteria apply.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2006-09; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (36):
- United States (36):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Springdale, Arkansas
  - Palo Alto, California
  - San Diego, California
  - New London, Connecticut
  - Bradenton, Florida
  - Miami, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Sandy Springs, Georgia
  - Savannah, Georgia
  - Smyrna, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Terre Haute, Indiana
  - Shreveport, Louisiana
  - Rockville, Maryland
  - Omaha, Nebraska
  - Cherry Hill, New Jersey
  - Brooklyn, New York
  - Minot, North Dakota
  - Beachwood, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Hilton Head Island, South Carolina
  - Austin, Texas
  - Houston, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Brown Deer, Wisconsin

REFERENCES:
- [Derived] Kornstein SG, Clayton AH, Bao W, Guico-Pabia CJ. A pooled analysis of the efficacy of desvenlafaxine for the treatment of major depressive disorder in perimenopausal and postmenopausal women. J Womens Health (Larchmt). 2015 Apr;24(4):281-90. doi: 10.1089/jwh.2014.4900. PMID 25860107
- [Derived] Kornstein SG, Jiang Q, Reddy S, Musgnung JJ, Guico-Pabia CJ. Short-term efficacy and safety of desvenlafaxine in a randomized, placebo-controlled study of perimenopausal and postmenopausal women with major depressive disorder. J Clin Psychiatry. 2010 Aug;71(8):1088-96. doi: 10.4088/JCP.10m06018blu. PMID 20797382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the United States from September 2006 to September 2007.
Pre-assignment Details: Patients were screened over 4 weeks.
Groups:
- Desvenlafaxine Succinate Sustained-Release (DVS SR): Double-blind Phase Days 1 to 7: 50 mg/day (one 50 mg tablet) Days 8 to 14: 100 mg/day (one 100 mg tables) Days 15 to 56: At the discretion of the investigator, patients assigned 100 mg/day (one 100 mg tablet) or 200 mg/day (two 100 mg tablets) Open-label Phase Days 57-63: 100 mg/day (one 100 mg tablet) Days 64-238: At the discretion of the investigator, patients assigned 100 mg/day (one 100 mg tablet) or 200 mg/day (two 100 mg tablets) Taper Phase Day 239 or at discontinuation: If patient taking 200 mg/day, then decreased to 100 mg for 7 days, and then decreased to 50 mg/day for 7 days. Patients taking 100 mg/day decreased to 50 mg/day for 7 days.
- Placebo: Double-blind Phase Placebo administered daily for 8 weeks Open-label Phase Days 57-63: 100 mg/day (one 100 mg tablet) Days 64-238: At the discretion of the investigator, patients assigned 100 mg/day (one 100 mg tablet) or 200 mg/day (two 100 mg tablets) Taper Phase Day 239 or at discontinuation: If patient taking 200 mg/day, then decreased to 100 mg/day for 7 days, and then decreased to 50 mg/day for 7 days. Patients taking 100 mg/day decreased to 50 mg/day for 7 days.
Period: Double-blind Phase
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Started | 256 | 125
Completed | 212 | 109
Not Completed | 44 | 16
Not completed — Adverse Event | 19 | 4
Not completed — Failed to return | 2 | 0
Not completed — Lost to Follow-up | 9 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Lack of Efficacy | 0 | 4
Not completed — Protocol deviation | 4 | 0
Period: Open-label Phase
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Started | 212 | 109
Completed | 155 | 79
Not Completed | 57 | 30
Not completed — Adverse Event | 19 | 7
Not completed — Failed to return | 4 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 5 | 3
Not completed — inadvertently reported study completers | 3 | 2
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Lack of Efficacy | 4 | 3
Not completed — Lack of continuance tolerability | 3 | 4
Not completed — did not take study drug | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo | Total
Number analyzed (Participants) | 256 | 125 | 381
Age Continuous [Mean (Standard Deviation); unit: years] | 52.01 (6.50) | 52.56 (7.17) | 52.19 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 256 | 125 | 381
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Psychiatric Rating Scale for Depression (HAM-D17) Score From Baseline to Week 8.
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2-4 scale (0=none/absent and 4=most severe) with a maximum total score of 50. Change= 8 week adjusted mean HAM-D17 minus baseline adjusted mean HAM-D17
Time Frame: Baseline to 8 weeks
Population: Double-blind phase; modified intent to treat population, which included all randomized patients with a baseline HAM-D17 score ≥18, who took ≥1 dose of study drug and had ≥1 post-baseline HAM-D17 evaluation. Mixed model repeated measures (MMRM) modeling included all available observed data for each patient and no missing values were imputed.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Number analyzed (Participants) | 157 | 81
units on scale | -12.64 (0.53) | -8.33 (0.74)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mixed Models Repeated Measures (MMRM) used baseline as a covariate and factors for center, week and treatment; Mean Difference (Final Values) = 4.32, 95% CI [2.53 to 6.11] — DVS SR adjusted mean change minus placebo adjusted mean change

2. Secondary Outcome: Percentage of Patients With Each Clinical Global Impression Improvement (CGI-I) Score
Description: CGI-I is a global rating scale that measures disease improvement. Using a 7-point scale, the clinician rates how much the patient's illness has improved or worsened relative to the baseline status (1= very much improved; 7= very much worse).
Time Frame: 8 weeks
Population: Double-blind phase, modified intent to treat population, which included all randomized patients with a baseline HAM-D17 score ≥18, took ≥1 dose of study drug and had ≥1 post-baseline HAM-D17 evaluation. Missing data handled by last observation carried forward (LOCF).
Measure: Number; unit: percentage of patients
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Number analyzed (Participants) | 186 | 97
percentage of patients
  1 (very much improved) | 42.5 | 22.7
  2 (much improved) | 25.3 | 18.6
  3 (minimally improved) | 16.7 | 17.5
  4 (no change) | 13.4 | 32.0
  5 (minimally worse) | 1.1 | 7.2
  6 (much worse) | 0.5 | 2.1
  7 (very much worse) | 0.5 | 0.0
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — DVS SR compared to Placebo for CGI-I scores of either 1 (very much improved) or 2 (much improved)

3. Secondary Outcome: Percentage of Patients Achieving Remission
Description: Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score of ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2-4 scale (0=none/absent and 4=most severe) with a maximum total score of 50.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Number analyzed (Participants) | 186 | 98
percentage of patients | 38.2 | 22.4
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Placebo; Test type: Superiority or Other; p = 0.008, Chi-squared — DVS SR compared with Placebo; Logistic regression model with treatment and site as factors and baseline score as a covariate; Odds Ratio (OR) = 2.132, 95% CI [1.22 to 3.74] — Adjusted odds ratio of DVS SR to Placebo. Odds ratio adjusted for baseline, treatment and site

4. Secondary Outcome: Percentage of Patients Achieving Response to Treatment
Description: A response is defined as ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2-4 scale (0=none/absent and 4=most severe) with a maximum total score of 50.
Time Frame: 8 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Number analyzed (Participants) | 186 | 98
percentage of patients | 58.6 | 31.6
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Placebo; Test type: Superiority or Other; p < 0.001, Chi-squared — DVS SR compared with Placebo; Logistic regression model with treatment and site as factors and baseline score as a covariate; Odds Ratio (OR) = 3.125, 95% CI [1.85 to 5.27] — Adjusted odds ratio of DVS SR to Placebo. Odd ratio adjusted for baseline, treatment and site

5. Secondary Outcome: Change in Hamilton Psychiatric Rating Scale for Anxiety (HAM-A) Score From Baseline to Week 8
Description: The HAM-A is a standardized, clinician-administered rating scale that assesses 14 items characteristically associated with major anxiety disorders. Items are scaled 0 - 4 (0=none and 4=very severe), with a maximum total score of 56. Change= 8 week adjusted mean HAM-A score minus baseline adjusted mean score.
Time Frame: Baseline to 8 weeks
Population: Double-blind phase; modified intent to treat population, which included all randomized patients with a baseline HAM-D17 score ≥18, took ≥1 dose of study drug and had ≥1 post-baseline HAM-D17 evaluation. Mixed model repeated measures (MMRM) modeling included all available observed data for each patient and no missing values were imputed.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Number analyzed (Participants) | 158 | 81
units on scale | -8.62 (0.44) | -5.89 (0.62)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Mixed model Repeated Measures (MMRM) analysis adjusted mean score for baseline score, time and center; Mean Difference (Net) = 2.74, 95% CI [1.24 to 4.23] — Adjusted mean difference = Placebo adjusted mean score minus DVS SR adjusted mean score

6. Secondary Outcome: Change in Dimension Health State EuroQol (EQ-5D) Score From Baseline to Week 8
Description: EQ-5D is a standardized, subject-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a single index value characterizing current health status using a 100-point visual analog scale (0=worst, 100=best). EQ-5D summary index is obtained with a formula that weights each level of the dimensions. The index-based score is interpreted along a continuum of 0 (death) to 1 (perfect health). Change=8 week score minus baseline score.
Time Frame: Baseline to 8 weeks
Population: Double-blind phase; modified intent to treat population, which included all randomized patients with a baseline HAM-D17 score ≥18, took ≥1 dose of study drug and had ≥1 post-baseline HAM-D17 evaluation.
Measure: Mean (Standard Error); unit: units on scale
Arm/Group | Desvenlafaxine Succinate Sustained-Release (DVS SR) | Placebo
Number analyzed (Participants) | 158 | 81
units on scale | 0.18 (0.02) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Desvenlafaxine Succinate Sustained-Release (DVS SR) vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Mixed Model Repeated Measures (MMRM) with treatment and site as factors and baseline as covariate; Mean Difference (Net) = -0.12, 95% CI [-0.18 to -0.06] — Adjusted mean difference = Placebo adjusted mean score minus DVS SR adjusted mean score

7. Secondary Outcome: Change in Hamilton Psychiatric Rating Scale for Depression (HAM-D17) Score From Open Label Baseline to 6 Months
Description: HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2-4 scale (0=none/absent and 4=most severe) with a maximum total s core of 50. Change= Final Evaluation mean HAM-D17 minus baseline mean HAM-D17.
Time Frame: open label baseline and 6 months
Population: Open-label phase safety population: All patients who completed the double-blind phase, elected to continue treatment in the open-label phase, and received at least 1 dose of study drug in the open-label phase. One patient did not have a baseline and at least 1 on therapy assessment.
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- DVS SR / DVS SR: Patients were in the DVS SR arm during both the double-blind and open-label phase.
- Placebo / DVS SR: Patients were in the Placebo arm during the double-blind phase and the DVS SR arm during the open-label phase.
Arm/Group | DVS SR / DVS SR | Placebo / DVS SR
Number analyzed (Participants) | 207 | 103
units on scale | -12.52 (7.17) | -12.45 (6.85)

8. Secondary Outcome: Clinical Global Impression Improvement (CGI-I) Score
Description: CGI-I is a global rating scale that measures disease improvement. Using a 7-point scale the clinician rates how much the patient's illness has improved or worsened relative to the baseline status (1= very much improved; 7= very much worse)
Time Frame: 6 months
Population: Open-label phase safety population: All patients who completed the double-blind phase, elected to continue treatment in the open-label phase, and received at least 1 dose of study drug in the open-label phase.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | DVS SR / DVS SR | Placebo / DVS SR
Number analyzed (Participants) | 208 | 103
units on scale | 1.55 (1.00) | 1.56 (0.99)

9. Secondary Outcome: Percentage of Patients Achieving Remission
Description: Remission is defined as a Hamilton Psychiatric Rating Scale for Depression (HAM-D17) score of ≤ 7. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2-4 scale (0=none/absent and 4=most severe) with a maximum total s core of 50.
Time Frame: 6 months
Population: as for outcome 7
Measure: Number; unit: percentage of patients
Arm/Group | DVS SR / DVS SR | Placebo / DVS SR
Number analyzed (Participants) | 207 | 103
percentage of patients | 55.6 | 48.5

10. Secondary Outcome: Percentage of Patients Achieving a Response to Treatment
Description: A responder is defined as a patient with ≥ 50% decrease from baseline on Hamilton Psychiatric Rating Scale for Depression - 17-item (HAM-D17) score. HAM-D17 is a standardized, clinician-administered rating scale that assesses 17 items characteristically associated with major depression. Items are scored on a 0 to 2-4 scale (0=none/absent and 4=most severe) with a maximum total score of 50.
Time Frame: 6 months
Population: as for outcome 7
Measure: Number; unit: percentage of patients responding
Arm/Group | DVS SR / DVS SR | Placebo / DVS SR
Number analyzed (Participants) | 207 | 103
percentage of patients responding | 70.5 | 66.0

11. Secondary Outcome: Change in Hamilton Psychiatric Rating Scale for Anxiety (HAM-A) Score From Open Label Baseline to 6 Months
Description: The HAM-A is a standardized, clinician-administered rating scale that assesses 14 items characteristically associated with major anxiety disorders. Items are scaled 0 - 4 (0=none and 4=very severe), with a maximum total score of 56. Change= Final Evaluation mean HAM-A score minus baseline mean score.
Time Frame: open label baseline to 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | DVS SR / DVS SR | Placebo / DVS SR
Number analyzed (Participants) | 207 | 103
units on scale | -10.95 (6.90) | -10.38 (5.64)

12. Secondary Outcome: Change in Dimension Health State EuroQol (EQ-5D) Score From Open Label Baseline to 6 Months
Description: as for outcome 6
Time Frame: open label baseline to 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | DVS SR / DVS SR | Placebo / DVS SR
Number analyzed (Participants) | 208 | 102
units on scale | 0.19 (0.26) | 0.22 (0.31)

13. Secondary Outcome: Discontinuation-Emergent Signs and Symptoms (DESS) Total Score
Description: DESS: a clinician-administered 43-item assessment that evaluates discontinuation-emergent symptoms resulting from the withdrawal from test article. The DESS total score is the sum of the number of "new symptoms" and "old (but worse) symptoms" (1) and 0 for "old and unchanged symptom," "absent," or "old symptom but improved" for a total possible range of 0 to 43. A higher score indicates more symptoms.
Time Frame: 6 months
Population: Open-label (OL) safety population: Patients completed double-blind and continued in OL with ≥1 dose study drug. Excluded patients lost to follow-up and discontinued with <4 wks therapy. Patients analyzed varied by time (0mg, 100mg, 200mg): Early Termination (n=9,98,207); Taper week 1 (n=4,76,193); Taper week 2 (n=5,75,195); Post-taper (n=5,71,192)
Measure: Mean (Standard Deviation); unit: units on scale
Groups:
- 0 mg: Placebo
- 100 mg: DVS SR 100mg dosage was reduced to DVS SR 50mg for 7 days.
- 200 mg: DVS SR 200mg dosage was reduced to DVS SR 100mg for 7 days and then further reduced to DVS SR 50mg from days 8 to 14.
Arm/Group | 0 mg | 100 mg | 200 mg
Number analyzed (Participants) | 9 | 98 | 207
units on scale
  End of 8 week DB / OL phase or early termination | 4.00 (5.05) | 2.07 (4.03) | 1.27 (3.40)
  Taper week 1 | 2.00 (2.16) | 3.32 (4.35) | 2.47 (3.61)
  Taper week 2 | 1.40 (3.13) | 5.29 (5.96) | 3.76 (4.71)
  Post-taper | 0.60 (0.89) | 1.41 (2.18) | 2.46 (3.97)
Statistical Analysis 1: Comparison: 0 mg vs 100 mg; 100mg vs. Placebo (0mg) post taper; Test type: Superiority or Other; p = 0.553, t-test, 2 sided — t-test adjusted by multiple comparison
Statistical Analysis 2: Comparison: 0 mg vs 200 mg; 200mg vs. Placebo (0mg) post taper; Test type: Superiority or Other; p = 0.034, t-test, 2 sided — t-test adjusted by multiple comparison

ADVERSE EVENTS:
Groups:
- Double-blind DVS SR: Days 1 to 7:
  Patients will be instructed to take 1-50mg tablet per day
  Days 8 to 14:
  Patients will be instructed to take 1-100mg tablet per day
  Days 15 to 56:
  At the discretion of the investigator, patients may be assigned to 100mg or 200mg tablets per day
- Double-blind Placebo: Placebo administered daily for 8 weeks
- Open-label DVS SR/ DVS SR: Patients were in the DVS SR arm during both the double-blind and open-label phase.
- Open-label Placebo/DVS SR: Patients were in the Placebo arm during the double-blind phase and the DVS SR arm during the open-label phase.
Arm/Group | Double-blind DVS SR | Double-blind Placebo | Open-label DVS SR/ DVS SR | Open-label Placebo/DVS SR
Serious Adverse Events (participants affected / at risk) | 3 | 2 | 12 | 2
Other Adverse Events (participants affected / at risk) | 217 | 94 | 198 | 97
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Double-blind DVS SR | Double-blind Placebo | Open-label DVS SR/ DVS SR | Open-label Placebo/DVS SR
Hypertension (Cardiac disorders) | 1/256 | 0/125 | 0/208 | 0/103
Skin carcinoma (Skin and subcutaneous tissue disorders) | 0/256 | 1/125 | 0/208 | 0/103
Psychotic depression (Nervous system disorders) | 1/256 | 0/125 | 0/208 | 0/103
Infection (General disorders) | 1/256 | 0/125 | 0/208 | 0/103
Cerebrovascular disorder (Cardiac disorders) | 0/256 | 1/125 | 0/208 | 0/103
Medication error (General disorders) | 1/256 | 0/125 | 0/208 | 0/103
Chest pain (General disorders) | 1/256 | 0/125 | 0/208 | 1/103
Uterine fibroids enlarged (Reproductive system and breast disorders) | 0/256 | 0/125 | 0/208 | 1/103
Accidental overdose (General disorders) | 0/256 | 0/125 | 3/208 | 0/103
Overdose (General disorders) | 0/256 | 0/125 | 2/208 | 0/103
Allergic reaction (General disorders) | 0/256 | 0/125 | 1/208 | 0/103
Cerebral ischemia (Vascular disorders) | 0/256 | 0/125 | 1/208 | 0/103
Supraventricular tachycardia (Cardiac disorders) | 0/256 | 0/125 | 1/208 | 0/103
Deep vein thrombosis (Vascular disorders) | 0/256 | 0/125 | 1/208 | 0/103
Coagulation disorder (Blood and lymphatic system disorders) | 0/256 | 0/125 | 1/208 | 0/103
Psychosis (Nervous system disorders) | 0/256 | 0/125 | 1/208 | 0/103
Skin melanoma (Skin and subcutaneous tissue disorders) | 0/256 | 0/125 | 1/208 | 0/103
Endometrial carcinoma (Reproductive system and breast disorders) | 0/256 | 0/125 | 1/208 | 0/103
Breast carcinoma (Reproductive system and breast disorders) | 0/256 | 0/125 | 1/208 | 0/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Double-blind DVS SR | Double-blind Placebo | Open-label DVS SR/ DVS SR | Open-label Placebo/DVS SR
Abdominal pain (General disorders) | 11/256 | 8/125 | 21/208 | 8/103
Asthenia (General disorders) | 17/256 | 10/125 | 21/208 | 11/103
Headache (General disorders) | 68/256 | 26/125 | 82/208 | 43/103
Infection (General disorders) | 16/256 | 10/125 | 40/208 | 18/103
Pain (General disorders) | 8/256 | 7/125 | 20/208 | 12/103
Hypertension (Vascular disorders) | 17/256 | 2/125 | 21/208 | 4/103
Vasodilatation (Vascular disorders) | 15/256 | 5/125 | 18/208 | 7/103
Anorexia (Gastrointestinal disorders) | 15/256 | 1/125 | 12/208 | 6/103
Constipation (Gastrointestinal disorders) | 36/256 | 8/125 | 37/208 | 22/103
Diarrhea (Gastrointestinal disorders) | 22/256 | 13/125 | 33/208 | 15/103
Dry mouth (Gastrointestinal disorders) | 61/256 | 12/125 | 56/208 | 23/103
Dyspepsia (Gastrointestinal disorders) | 16/256 | 2/125 | 20/208 | 4/103
Nausea (Gastrointestinal disorders) | 43/256 | 15/125 | 52/208 | 32/103
Dizziness (Nervous system disorders) | 29/256 | 9/125 | 6/208 | 6/103
Insomnia (Nervous system disorders) | 29/256 | 8/125 | 32/208 | 16/103
Nervousness (Nervous system disorders) | 13/256 | 4/125 | 14/208 | 7/103
Somnolence (Nervous system disorders) | 37/256 | 9/125 | 27/208 | 15/103
Sweating (Skin and subcutaneous tissue disorders) | 17/256 | 3/125 | 20/208 | 12/103
Accidental injury (General disorders) | 0/256 | 0/125 | 35/208 | 12/103
Back pain (General disorders) | 0/256 | 0/125 | 13/208 | 6/103
Flu syndrome (General disorders) | 0/256 | 0/125 | 11/208 | 5/103
Vomiting (Gastrointestinal disorders) | 0/256 | 0/125 | 7/208 | 9/103
Weight gain (Metabolism and nutrition disorders) | 0/256 | 0/125 | 17/208 | 9/103
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/256 | 0/125 | 18/208 | 6/103
Abnormal dreams (Nervous system disorders) | 0/256 | 0/125 | 15/208 | 1/103
Anxiety (Nervous system disorders) | 0/256 | 0/125 | 6/208 | 6/103
Hostility (Nervous system disorders) | 0/256 | 0/125 | 3/208 | 7/103
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0/256 | 0/125 | 12/208 | 10/103
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0/256 | 0/125 | 14/208 | 7/103
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0/256 | 0/125 | 23/208 | 11/103
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0/256 | 0/125 | 19/208 | 9/103
Abnormal vision (Eye disorders) | 0/256 | 0/125 | 13/208 | 5/103
Tinnitus (Ear and labyrinth disorders) | 0/256 | 0/125 | 15/208 | 2/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.